CLINICAL TRIAL: NCT04313881
Title: ENHANCE: A Randomized, Double-blind, Multicenter Study Comparing Magrolimab in Combination With Azacitidine Versus Azacitidine Plus Placebo in Treatment-naïve Patients With Higher Risk Myelodysplastic Syndrome
Brief Title: Magrolimab + Azacitidine Versus Azacitidine + Placebo in Untreated Participants With Myelodysplastic Syndrome (MDS)
Acronym: ENHANCE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study discontinued due to futility based on a planned analysis
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5F9009; 2020-004287-26 (EudraCT Number)
Record Dates: First submitted 2020-03-11; First posted 2020-03-18 (Actual); Results first posted 2024-03-21 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — magrolimab; Azacitidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Magrolimab + Azacitidine (Experimental): Participants will receive the following magrolimab and azacitidine dosing regimens:
  Magrolimab:
  Magrolimab Priming Dose:
  * 1 mg/kg on Days 1 and 4
  * 15 mg/kg on Day 8
  * 30 mg/kg on Days 11, 15, followed by weekly administration for 5 doses (on Days 22, 29, 36, 43, and 50)
  Magrolimab Maintenance Dose:
  * 30 mg/kg on Day 57 and 30 mg/kg every 2 weeks thereafter.
  Azacitidine: 75 mg/m^2 on Days 1 to 7 (or Days 1 to 5 and 8 to 9) of each 28-day cycle.
  Interventions: Drug: Magrolimab; Drug: Azacitidine
- Control Arm (Placebo + Azacitidine) (Placebo Comparator): Participants will receive the following placebo dosing regimens to mirror magrolimab dosing regimen in addition to azacitidine:
  Placebo: On Days 1 and 4; Day 8; Days 11, 15, followed by weekly administration for 5 doses (on Days 22, 29, 36, 43, and 50). Additionally, placebo was administered on Day 57 and every 2 weeks thereafter.
  Azacitidine: 75 mg/m^2 on Days 1 to 7 (or Days 1 to 5 and 8 to 9) of each cycle.
  Interventions: Drug: Azacitidine; Drug: Placebo

INTERVENTIONS:
Drug: Magrolimab — Administered intravenously
  Other Names: Hu5F9-G4; GS-4721
  Arms: Magrolimab + Azacitidine
Drug: Azacitidine — Administered either subcutaneously (SC) or intravenously (IV) according to region-specific drug labeling
Drug: Placebo — Placebo to match magrolimab administered intravenously
  Arms: Control Arm (Placebo + Azacitidine)

SUMMARY:
The primary objective of this study is to evaluate the efficacy of magrolimab in combination with azacitidine compared to that of azacitidine plus placebo in previously untreated participants with intermediate/high/very high risk myelodysplastic syndrome (MDS) by Revised International Prognostic Scoring System (IPSS-R) as measured by complete remission (CR) and overall survival (OS).

ELIGIBILITY:
Key Inclusion Criteria:

* Participants with Myelodysplastic Syndrome (MDS) defined according to World Health Organization classification, with Revised International Prognostic Scoring System (IPSS-R) prognostic risk category of intermediate, high, or very high risk.
* Adequate performance status and hematological, liver, and kidney function.

Key Exclusion Criteria:

* Immediate eligibility for allogenic stem cell transplant (SCT), as determined by the investigator, with an available donor.
* Prior treatment with Cluster of Differentiation (CD) 47 or Signal-regulatory protein alpha (SIRPα)-targeting agents.
* Any prior antileukemic therapy for treatment of intermediate, high, very high risk MDS per IPSS-R.
* Second malignancy, except treated basal cell or localized squamous skin carcinomas, localized prostate cancer, or other malignancies for which participants are not on active anticancer therapies and have had no evidence of active malignancy for at least ≥ 1 year.
* Contraindications to azacitidine.
* Clinical suspicion of active central nervous system (CNS) involvement by MDS.
* Known active or chronic hepatitis B or C infection or human immunodeficiency virus in medical history .
* Active hepatitis B virus and/or active hepatitis C virus, and/or HIV following testing at screening.
* Pregnancy or active breastfeeding.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 539 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (169):
- United States (47):
  - University of Alabama Birmingham, Birmingham, Alabama
  - University of Arkansas for Medical Sciences IRB, Little Rock, Arkansas
  - City of Hope, Duarte, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - UCLA Ronald Reagan Medical Center, Los Angeles, California
  - UC Irvine Health, Orange, California
  - Stanford Cancer Institute, Palo Alto, California
  - University of California, Davis Comprehensive Cancer Center, Sacramento, California
  - University of Miami Hospital and Clinics / Sylvester Comprehensive Cancer Center, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - The University of Chicago Medical Center, Chicago, Illinois
  - University of Kansas Clinical Research Center, Fairway, Kansas
  - Tulane Medical Center, New Orleans, Louisiana
  - University of Maryland, Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Johns Hopkins Medicine - The Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute (DFCI), Boston, Massachusetts
  - University of Michigan Medical School, Ann Arbor, Michigan
  - University of Minnesota Medical Center, Fairview, Minneapolis, Minnesota
  - Mid America Division, Inc., Kansas City, Missouri
  - Washington University School of Medicine - Siteman Cancer Center, St Louis, Missouri
  - Roswell Park Cancer Institute, Buffalo, New York
  - Weill Cornell Medicine-New York Presbyterian Hospital, New York, New York
  - Mount Sinai Health System, New York, New York
  - Columbia University Medical Center - Herbert Irving Pavilion, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - DUHS Duke Cancer Center, Durham, North Carolina
  - The Ohio State University Wexner Medical Center / James Cancer Hospital, Columbus, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health & Science University Pharmacy Services, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University, Sidney Kimmel Cancer Center; Clinical Research Organization, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Prisma Health Cancer Center, Greenville, South Carolina
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - Texas Oncology - Baylor Charles A. Simmons Cancer Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - Seattle Cancer Care Alliance, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Froedtert Hospital & the Medical College of Wisconsin, Milwaukee, Wisconsin
- Australia (16):
  - Gosford Hospital, Gosford, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Icon Cancer Foundation, South Brisbane, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Center, Bedford Park, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Eastern Health, Box Hill, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - Peninsula Private Hospital, Frankston, Victoria
  - Barwon Health, University Hospital Geelong, Geelong, Victoria
  - Cabrini Hospital Malvern, Malvern, Victoria
  - The Alfred Hospital, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Austria (2):
  - Uniklinikum Salzburg, Salzburg
  - Hanusch kranhenkaus, 3. Medizinische Abteilung, Vienna
- Belgium (7):
  - ZNA Middelheim, Antwerp
  - ULB Hopital Erasme, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - UZ Brussel, Brussels
  - Chu Ucl Namur Site Godinne, Godinne
  - UZ Leuven, Leuven
  - AZ Turnhout, Campus St. Elisabeth, Turnhout
- Canada (4):
  - Tom Baker Cancer Centre, Calgary
  - QEII Health Sciences Centre, Halifax
  - Eastern Regional Health Authority, St. John's
  - University Health Network, Toronto
- Czechia (2):
  - Fakultni nemocnice Olomouc, Hemato-onkologicka klinika, Olomouc
  - Fakultni nemocnice Ostrava, Klinika hemato-onkologicka, Ostrava
- Finland (2):
  - Helsinki University Central Hospital, Helsinki
  - Oulu University Hospital, Oulu
- France (13):
  - CHU Amiens-Picardie, Amiens
  - Hopital Henri Mondor, Créteil
  - CHU de Grenoble Alpes, La Tronche
  - Institut Paoli Calmettes, Marseille
  - Hopital Saint Eloi, Montpellier
  - CHU de Nantes, Nantes
  - CHU de Nice-l Archet, Nice
  - Hopital Saint Louis, Paris
  - Institut Gustave Roussy, Paris
  - Hopital Haut-Leveque, Pessac
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU de Poitiers - Hopital de la Miletrie, Poitiers
  - CHU de Rennes- Hopital Pontchaillou, Rennes
- Germany (6):
  - Universitatsmedizin der Johannes Gutenberg Universitat Mainz, III. Medizinische Klinik und Poliklinik, Braunschweig
  - Universitatsklinikum Carl Gustav Carus, Dresden
  - Marien hospital, klinik fur onkologie, hamatologie und palliavmedizin, Düsseldorf
  - Universitatsklinikum Essen, Essen
  - Universitat Leipzig, Leipzig
  - Robert-Bosch-Krankenhaus, GmBH, Hamatologie, Onkologie und Palliativmedizin, Stuttgart
- Hong Kong (5):
  - Hong Kong Sanatorium & Hospital, Hong Kong
  - Princess Margaret Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - The Chinese University of Hong Kong, Prince of Wales Hospital, Hong Kong
  - Tuen Mun Hospital, Hong Kong
- Hungary (8):
  - Semmelweis Egyetem Belgyógyászati és Hematológiai Kilnika, Budapest
  - Debreceni Egyetem Klinikai Központ, Debrecen
  - Petz Aladar Egyetemi Oktato Korhaz II. Belgyogyaszat - Hematologial Osztaly, Győr
  - Kaposi Mor Teaching Hospital, Kaposvár
  - Bács-Kiskun Megyei Kórház, Kecskemét
  - SzSzB Megyei Korhazak es Egyetemi Oktatokorhaz, Nyíregyháza
  - University of Pecs, Pécs
  - Szent Borbála Hospital, Tatabánya
- Italy (9):
  - SC Ematologica- Azienda Ospedaliera Nazionale SS. Antonio e Biagio e C. Arrigo, Alessandria
  - U.O Ematologica- ASST degli Spedali Civili di Brescia, Brescia
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - U.O.C Ematologia - Dipartimento di Medicina Interna, Fondazione IRCCS Ca'Granda Ospedale Maggiore Policlinico, Milan
  - U.O di Ematologia, Ospedale San Gerardo- ASST Monza, Monza
  - S. C. Ematologia Azienda Ospedaliero - Universitaria Maggiore Della Carita, Novara
  - Azienda Ospedaliera Ospedali Riuniti Marche Nord, Pesaro
  - SC di Oncoematologia - Azienda Ospedaliera Santa Maria, Terni
  - SC Ematologica, ASST Sette Laghi, Ospedale di Circolo e Fondazione Macchi, Varese
- Netherlands (2):
  - University Medical Center Groningen, Groningen
  - Medisch Centrum Leeuwarden, Leeuwarden
- New Zealand (5):
  - Christchurch Hospital, Christchurch
  - Southern District Health Board, Dunedin
  - Auckland City Hospital, Grafton
  - Waikato Hospital, Hamilton
  - Midcentral District Health Board, Palmerston North
- Norway (4):
  - Haukeland Universitetssjukehus, seksjon for blodsjukdommar- klinisk studieteam, Bergen
  - Akershus University Hospital, Loerenskog
  - Oslo University Hospital, Oslo
  - Stavanger universitetssjukehus, Stavanger
- Poland (3):
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Szpital Uniwersytecki w Krakowie, Oddzial Kliniczny Hematologii, Krakow
  - Centrum Onkologii Ziemi Lubelskiej im. św. Jana z Dukli, Lublin
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wroclawiu, Wroclaw
- Portugal (6):
  - Centro Clinico Academico de Braga, Hospital de Braga, E.P.E, Braga
  - Champalimaud Foundation, Lisbon
  - Hospital da Luz, Lisbon
  - Centro Hospitalar Universitario Sao Joao. E.P.E, Porto
  - Instituto Portugues de Oncologia do Porto Francisco Gentil, EPE, Porto
  - Centro Hospitalar Vila Nova de Gaia/Espinho, Porto
- Spain (15):
  - Area Sanitaria de Santiago de Compostela y Barbanza. Complejo Hospitalario Universitario de SantiagoD, A Coruña
  - OSI Araba, Hospital Universitario de Alava, Hospital Txagorritxu, Alava
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Institut Catala d'Oncologia Girona, Girona
  - Institut Catala d'Oncologia, Hospital Duran i Reynals, L'Hospitalet de Llobregat
  - MD Anderson Cancer Center Madrid, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario La Paz, Edificio General, 6 Planta. Despacho de Hematologia, Madrid
  - Hospital Universitario Quironsalud Madrid. Servico de Hematologica y Hemoterapia, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Centro Hospitalar Universitario Sao Joao, Pamplona
  - Complejo Asistencial Universitario de Salamanca- Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
- Switzerland (3):
  - Istituto Oncologico Della Svizzera Italiana- IOSI, EOC, Clinica di Ematologia, Bellinzona
  - University of Bern, Bern
  - Universitaetsspital Zurich - Klinik fur Medizinische Onkologie und Hematologie, Zurich
- Turkey (Türkiye) (6):
  - Hematoloji Bilim Dali, Yenimahalle, Ankara
  - Gazi Universitesi Tip Fakultesi, Ankara
  - Ankara Universitesi Tip Fakultesi Cebeci Hastanesi, Ankara
  - Dokuz Eylul Universitesi Tip Fakultesi Onkoloji Enstitusu, Inciralt
  - Mersin University Medical, Mersin
  - Tekirdag Namik Kemal Universitesi Tip Fakultesi, Tekirdağ
- United Kingdom (4):
  - University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - United Lincolnshire Hospital NHS Trust, Boston
  - Kent and Canterbury Hospital- East Kent Hospitals University NHS Foundation Trust, Canterbury
  - Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sallman DA, Al Malki MM, Asch AS, Wang ES, Jurcic JG, Bradley TJ, Flinn IW, Pollyea DA, Kambhampati S, Tanaka TN, Zeidner JF, Garcia-Manero G, Jeyakumar D, Komrokji R, Lancet J, Kantarjian HM, Gu L, Zhang Y, Tan A, Chao M, O'Hear C, Ramsingh G, Lal I, Vyas P, Daver NG. Magrolimab in Combination With Azacitidine in Patients With Higher-Risk Myelodysplastic Syndromes: Final Results of a Phase Ib Study. J Clin Oncol. 2023 May 20;41(15):2815-2826. doi: 10.1200/JCO.22.01794. Epub 2023 Mar 8. PMID 36888930
- See also: Gilead Clinical Trials Website — https://www.gileadclinicaltrials.com/study/?id=5F9009

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in North America, Asia-Pacific Region, and Europe.
Pre-assignment Details: 854 participants were screened.
Groups:
- Magrolimab + Azacitidine: Participants received the following magrolimab and azacitidine dosing regimens:
  Magrolimab was administered as an intravenous (IV) priming dose of 1 mg/kg on Days 1 and 4; 15 mg/kg on Day 8; 30 mg/kg on Days 11, 15, followed by weekly administration for 5 doses (on Days 22, 29, 36, 43, and 50). Following priming dose, magrolimab maintenance dose of 30 mg/kg was administered on Day 57 and 30 mg/kg every 2 weeks thereafter.
  Azacitidine 75 mg/m^2 was administered either subcutaneously (SC) or IV on Days 1 to 7 (or Days 1 to 5 and 8 to 9) of each 28-day cycle.
  The maximum duration of treatment was up to approximately 2.6 years.
- Placebo + Azacitidine: Participants received the following placebo dosing regimens to mirror magrolimab dosing regimen in addition to azacitidine:
  Placebo was administered as an IV on Days 1 and 4; Day 8; Days 11, 15, followed by weekly administration for 5 doses (on Days 22, 29, 36, 43, and 50). Additionally, placebo was administered on Day 57 and every 2 weeks thereafter.
  Azacitidine 75 mg/m^2 was administered either subcutaneously (SC) or IV on Days 1 to 7 (or Days 1 to 5 and 8 to 9) of each 28-day cycle.
  The maximum duration of treatment was up to approximately 2.5 years.
Period: Overall Study
Arm/Group | Magrolimab + Azacitidine | Placebo + Azacitidine
Started | 268 | 271
Completed | 0 | 0
Not Completed | 268 | 271
Not completed — Death | 138 | 126
Not completed — Study terminated by sponsor | 108 | 129
Not completed — Consent withdrawn | 19 | 15
Not completed — Reason not Specified | 3 | 1

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat (ITT) Analysis Set included all participants who were randomized in the study, with treatment assignments designated according to the treatment that participants were randomized to.
Groups:
- Total: Total of all reporting groups
Arm/Group | Magrolimab + Azacitidine | Placebo + Azacitidine | Total
Number analyzed (Participants) | 268 | 271 | 539
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 64 | 81 | 145
  >=65 years | 204 | 190 | 394
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (9.2) | 68 (9.8) | 69 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 94 | 181
  Male | 181 | 177 | 358
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 21 | 34
  Non Hispanic or Latino | 227 | 219 | 446
  Unknown | 5 | 7 | 12
  Not Reported / Missing | 23 | 24 | 47
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian Or Alaska Native | 0 | 0 | 0
  Asian | 14 | 14 | 28
  Black or African American | 11 | 9 | 20
  Native Hawaiian Or Other Pacific Islander | 0 | 0 | 0
  White | 209 | 207 | 416
  Multiple | 1 | 0 | 1
  Not reported / Missing | 33 | 41 | 74
Region of Enrollment [Count of Participants; unit: Participants]
  Hong Kong | 5 | 3 | 8
  Hungary | 0 | 1 | 1
  United States | 175 | 177 | 352
  United Kingdom | 6 | 3 | 9
  Switzerland | 0 | 2 | 2
  Portugal | 2 | 1 | 3
  Spain | 11 | 16 | 27
  New Zealand | 1 | 5 | 6
  Canada | 0 | 2 | 2
  Turkey | 1 | 1 | 2
  Belgium | 1 | 0 | 1
  Norway | 1 | 0 | 1
  Finland | 0 | 2 | 2
  Poland | 3 | 7 | 10
  Italy | 11 | 2 | 13
  France | 9 | 12 | 21
  Australia | 40 | 35 | 75
  Germany | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Remission (CR)
Description: The percentage of participants (CR rate) are participants who reach morphologic CR (morphological blast of ≤ 5% and recovery of absolute neutrophil count (ANC), platelets, and hemoglobin from complete blood counts as well as peripheral blast) based on Investigator-assessed International Working Group (IWG) myelodysplastic syndrome (MDS) criteria on or prior to initiation of any new anticancer therapy, including stem cell therapy (SCT). Percentages were rounded off.
Time Frame: From randomization up to 31.01 months
Population: Participants from intent-to-treat analysis set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Magrolimab + Azacitidine | Placebo + Azacitidine
Number analyzed (Participants) | 268 | 271
percentage of participants | 21.3 [16.5 to 26.7] | 23.6 [18.7 to 29.1]
Statistical Analysis 1: Comparison: Magrolimab + Azacitidine vs Placebo + Azacitidine; Test type: Superiority; p = 0.5218, Cochran-Mantel-Haenszel — 2-sided P-value, odds ratio and its 95% CI were based on Cochran-Mantel-Haenszel (CMH) method stratified by stratification factors (geographic region, cytogenetic risk status, and bone marrow blast percentage); Odds Ratio (OR) = 0.876, 95% CI 2-sided [0.585 to 1.312]

2. Primary Outcome: Overall Survival (OS)
Description: OS is defined as the number of months measured from the date of randomization to the date of death from any cause. Kaplan Meier (KM) estimates were used for analysis.
Time Frame: From randomization up to 32.62 months
Population: Participants from intent-to-treat analysis set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Magrolimab + Azacitidine | Placebo + Azacitidine
Number analyzed (Participants) | 268 | 271
months | 15.9 [13.3 to 19.5] | 18.6 [14.9 to 26.2]
Statistical Analysis 1: Comparison: Magrolimab + Azacitidine vs Placebo + Azacitidine; Test type: Superiority; p = 0.1299, Log Rank — 2-sided P-value was based on stratified log-rank test, stratified by stratification factors; Hazard Ratio (HR) = 1.203, 95% CI 2-sided [0.947 to 1.528] — Hazard ratio and its 95% confidence interval (CI) were calculated using the Cox proportional hazards regression model, stratified by stratification factors

3. Secondary Outcome: Duration of CR (DOCR)
Description: DOCR=Time from first CR date to the first date of relapse, disease progression (PD) or death, prior to initiation of any new anticancer therapy excluding SCT whichever occurs earlier. PD is defined as: <5% blasts: ≥50 increase in blasts to >5% blasts,5%-10% blasts: ≥50% increase in blasts to >10% blasts, 10%-20% blasts: ≥50% increase in blasts to >20% blasts,20%-30% blasts: ≥50% increase in blasts to >30% blasts, any of the following: at least 50% decrement from maximum remission/response in granulocytes or platelets. Reduction in Hgb by ≥2 g/dL / Transfusion dependence. Relapse is defined as return to pretreatment bone marrow blast percentage / decrement of ≥ 50% from maximum remission/response levels in granulocytes or platelets/ reduction in Hgb concentration by ≥ 1.5 g/dL or transfusion dependence. CR is defined in outcome measure 1. KM estimates were used for analysis.
Time Frame: From randomization up to 31.01 months
Population: Participants from intent-to-treat analysis set who achieved CR were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Magrolimab + Azacitidine | Placebo + Azacitidine
Number analyzed (Participants) | 57 | 64
months | 10.9 [8.9 to 16.7] | 11.1 [8.1 to NA] — Upper limit of CI was not estimable due to low number of participants with events.

4. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants who reach objective response including CR, partial remission (PR), marrow CR or hematological improvement prior to initiation of any new anticancer therapy including SCT for MDS per IWG 2006 criteria per investigator's evaluation. CR is defined in outcome measure 1.
  PR is defined as all CR criteria if abnormal before treatment except, one marrow blasts decreased by ≥ 50% over pretreatment but still > 5% cellularity and morphology not relevant.
  Marrow CR is defined as bone marrow ≤ 5% myeloblasts and decrease by ≥ 50% over pretreatment, stable disease with any hematological improvement, peripheral blood: if hematological improvement responses, they were noted in addition to marrow CR.
  Stable Disease: Failure to achieve at least PR, but no evidence of progression for > 8 weeks.
  Percentages were rounded off.
Time Frame: From randomization up to 31.01 months
Population: Participants from intent-to-treat analysis set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Magrolimab + Azacitidine | Placebo + Azacitidine
Number analyzed (Participants) | 268 | 271
percentage of participants | 53.7 [47.6 to 59.8] | 58.7 [52.6 to 64.6]
Statistical Analysis 1: Comparison: Magrolimab + Azacitidine vs Placebo + Azacitidine; Test type: Superiority; p = 0.2563, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.821, 95% CI 2-sided [0.584 to 1.155]

5. Secondary Outcome: Duration of Response (DOR)
Description: DOR is measured from time measurement criteria are first met for objective response to first date of relapse, disease progression (PD) /death, prior to initiation of any new anticancer therapy excluding SCT whichever occurs earlier.
  Disease progression and relapse have been defined in outcome measure number 3. KM estimates were used for analysis.
Time Frame: From randomization up to 31.01 months
Population: Participants from intent-to-treat analysis set with objective response were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Magrolimab + Azacitidine | Placebo + Azacitidine
Number analyzed (Participants) | 144 | 159
months | 10.1 [8.1 to 12.5] | 10.2 [7.6 to 12.9]

6. Secondary Outcome: Red Blood Cell (RBC) Transfusion Independence Rate
Description: RBC transfusion independence rate is defined as the percentage of participants who have a 56-day or longer period with no RBC transfusions at any time between randomization and initiation of any new anticancer therapy, including SCT, among all participants who were RBC transfusion-dependent at Baseline. Percentages were rounded off.
Time Frame: From randomization up to 31.01 months
Population: Participants from intent-to-treat analysis set who were RBC transfusion-dependent at baseline were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Magrolimab + Azacitidine | Placebo + Azacitidine
Number analyzed (Participants) | 140 | 125
percentage of participants | 27.9 [20.6 to 36.1] | 35.2 [26.9 to 44.2]
Statistical Analysis 1: Comparison: Magrolimab + Azacitidine vs Placebo + Azacitidine; Test type: Superiority; p = 0.2191, Cochran-Mantel-Haenszel — 95% CI for transfusion independence rate was based on Clopper-Pearson exact method. 2-sided P-value, odds ratio and its 95% CI were based on Cochran-Mantel-Haenszel (CMH) method stratified by stratification factors; Odds Ratio (OR) = 0.720, 95% CI 2-sided [0.427 to 1.212]

7. Secondary Outcome: Event Free Survival (EFS)
Description: EFS is defined as the time from randomization to transformation to acute myeloid leukemia (AML) or death from any cause, whichever occurs first.
  Transformation assessments and deaths post SCT were included in the analysis. KM estimates were used for analysis
Time Frame: From randomization up to 31.01 months
Population: Participants from intent-to-treat analysis set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Magrolimab + Azacitidine | Placebo + Azacitidine
Number analyzed (Participants) | 268 | 271
months | 13.0 [10.2 to 15.9] | 12.9 [10.8 to 14.6]
Statistical Analysis 1: Comparison: Magrolimab + Azacitidine vs Placebo + Azacitidine; Test type: Superiority; p = 0.8788, Log Rank — 2-sided P-value was based on stratified log-rank test, stratified by stratification factors; Hazard Ratio (HR) = 0.979, 95% CI 2-sided [0.746 to 1.285] — Hazard ratio and its 95% CI were calculated using the Cox proportional hazards regression model, stratified by stratification factors

8. Secondary Outcome: Percentage of Participants With CR in Participants With TP53 Mutation
Description: CR in TP53 mutant population is defined as the percentage of participants who achieve a morphologic CR based on investigator assessments using IWG criteria on or prior to initiation of any new anticancer therapy, including SCT in TP53 mutant population. Percentages were rounded off.
Time Frame: From randomization up to 31.01 months
Population: Participants from intent-to-treat analysis set with TP53 mutation were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Magrolimab + Azacitidine | Placebo + Azacitidine
Number analyzed (Participants) | 79 | 64
percentage of participants | 17.7 [10.0 to 27.9] | 32.8 [21.6 to 45.7]
Statistical Analysis 1: Comparison: Magrolimab + Azacitidine vs Placebo + Azacitidine; Test type: Superiority; p = 0.0375, Cochran-Mantel-Haenszel — 2-sided P-value, odds ratio and its 95% CI were based on unstratified Cochran-Mantel-Haenszel (CMH) method; Odds Ratio (OR) = 0.441, 95% CI 2-sided [0.203 to 0.960] — 95% CI for response rate was based on Clopper-Pearson exact method

9. Secondary Outcome: Minimal Residual Disease (MRD)-Negative Response Rate
Description: The MRD-negative response rate is defined as the percentage of participants who achieved a morphologic CR or marrow CR based on Investigator-assessed IWG criteria and reached MRD-negative disease status prior to initiation of any new anticancer therapy, including SCT. MRD-negative disease status was assessed using a multiparameter flow cytometry-based assay performed by a central laboratory.
  Morphologic CR and marrow CR are defined in outcome measures 1 and 4, respectively.
  Percentages were rounded off.
Time Frame: From randomization up to 31.01 months
Population: Participants from intent-to-treat analysis set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo + Azacitidine: Participants received the following placebo dosing regimens to mirror magrolimab dosing regimen in addition to azacitidine:
  Placebo was administered IV on Days 1 and 4; Day 8; Days 11, 15, followed by weekly administration for 5 doses (on Days 22, 29, 36, 43, and 50). Additionally, placebo was administered on Day 57 and every 2 weeks thereafter.
  Azacitidine 75 mg/m^2 was administered either subcutaneously (SC) or IV on Days 1 to 7 (or Days 1 to 5 and 8 to 9) of each 28-day cycle.
  The maximum duration of treatment was up to approximately 2.5 years.
Arm/Group | Magrolimab + Azacitidine | Placebo + Azacitidine
Number analyzed (Participants) | 268 | 271
percentage of participants | 21.6 [16.9 to 27.1] | 22.5 [17.7 to 28.0]
Statistical Analysis 1: Comparison: Magrolimab + Azacitidine vs Placebo + Azacitidine; Test type: Superiority; p = 0.7950, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.947, 95% CI 2-sided [0.629 to 1.426] — 95% CI for response rate was based on Clopper-Pearson exact method

10. Secondary Outcome: Time to Transformation to AML
Description: Time to transformation to AML is defined as the time from randomization to the collection date of bone marrow sample leading to documented AML diagnosis. Transformation assessments post SCT were included in the analysis.KM estimates were used for analysis.
Time Frame: From randomization up to 31.01 months
Population: Participants from intent-to-treat analysis set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Magrolimab + Azacitidine | Placebo + Azacitidine
Number analyzed (Participants) | 268 | 271
months | NA [21.2 to NA] — Median and upper limit of CI was not estimable due to low number of participants with events. | 25.5 [25.5 to NA] — Upper limit of CI was not estimable due to low number of participants with events.
Statistical Analysis 1: Comparison: Magrolimab + Azacitidine vs Placebo + Azacitidine; Test type: Superiority; p = 0.4610, Log Rank — 2-sided P-value was based on stratified log-rank test, stratified by stratification factors; Hazard Ratio (HR) = 0.837, 95% CI 2-sided [0.522 to 1.343] — [estimate comment as in outcome 7, analysis 1]

11. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from randomization to the date of documented DP (including treatment failure by IWG criteria or relapse after PR/CR), or death from any cause, whichever occurs first. Response assessments and deaths post SCT were included in the analysis. Treatment failure is defined as, Death during treatment or disease progression characterized by worsening cytopenia, increase in percentage of bone marrow blasts, or progression to a more advanced MDS FAB subtype than pretreatment. Relapse after CR or PR = Return to pretreatment bone marrow blast percentage / Decrement of ≥ 50% from maximum remission/response levels in granulocytes or platelets / Reduction in Hgb concentration by ≥ 1.5 g/dL or transfusion dependence.
  CR, PR and PD are defined in outcome measures 1, 4 and 5 respectively. KM estimates were used for analysis.
Time Frame: From randomization up to 31.01 months
Population: Participants from intent-to-treat analysis set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Magrolimab + Azacitidine | Placebo + Azacitidine
Number analyzed (Participants) | 268 | 271
months | 9.0 [8.3 to 10.9] | 9.4 [8.6 to 11.4]
Statistical Analysis 1: Comparison: Magrolimab + Azacitidine vs Placebo + Azacitidine; Test type: Superiority; p = 0.8720, Log Rank — 2-sided P-value was based on stratified log-rank test, stratified by stratification factors (geographic region, cytogenetic risk status, and bone marrow blast percentage); Hazard Ratio (HR) = 1.020, 95% CI 2-sided [0.802 to 1.297] — [estimate comment as in outcome 7, analysis 1]

12. Secondary Outcome: Functional Assessment of Cancer Therapy-Anemia (FACT-Anemia) Response Rate
Description: The FACT-Anemia response rate is defined as the percentage of participants who showed clinically meaningful improvement in health-related quality of life (HRQoL) based on the score from the FACT-Anemia instrument prior to initiation of any new anticancer therapy, including SCT. The minimal clinically meaningful difference of 7.0 was used as cutoff for clinically meaningful improvement.
  The FACT-Anemia instrument consists of 5 subscales, including physical well-being, emotional well-being, functional well-being, social well-being, and anemia symptoms. Each subscale measures items on a 5-point Likert scale from 0 to 4, where 0 = not at all and 4 = very much. The subscales are scored by summing points from all questions, then converting this sum to a 100 point scale; 0 indicates the poorest quality of life (QOL) and 100 denotes the highest QOL.
  Percentages were rounded off.
Time Frame: Up to week 136
Population: Participants from intent-to-treat analysis set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Magrolimab + Azacitidine | Placebo + Azacitidine
Number analyzed (Participants) | 268 | 271
percentage of participants | 37.7 [31.9 to 43.8] | 49.8 [43.7 to 55.9]
Statistical Analysis 1: Comparison: Magrolimab + Azacitidine vs Placebo + Azacitidine; Test type: Superiority — 2-sided P-value, odds ratio and its 95% CI were based on Cochran-Mantel-Haenszel (CMH) method stratified by stratification factors; p = 0.0048, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.605, 95% CI 2-sided [0.428 to 0.857] — 95% CI for response rate was based on Clopper-Pearson exact method

13. Secondary Outcome: Percentage of Participants Experiencing Treatment-Emergent Adverse Events (TEAE)
Description: TEAE's are defined as any AEs with an onset date on or after the study drug start date, no later than 70 days after study drug last dose date or day before initiation of new anticancer therapy including SCT. If AE onset date is on or before last dose date, it is considered as TEAE regardless of start of new anticancer therapy. An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with use of an investigational product or other protocol imposed intervention, regardless of attribution. An event is considered "serious", if it results death, life-threatening, inpatient or prolongation hospitalization, incapacity or substantial disruption of the ability to conduct normal functions, a congenital anomaly/birth defect, and important medical events.
Time Frame: First dose date up to 135.9 weeks plus 70 days (Up to 2.8 years)
Population: Participants from safety analysis set with data available were analyzed. The safety analysis set included all randomized participants who took at least 1 dose of any study treatment, with treatment assignment designated according to the actual treatment received.
Measure: Number; unit: percentage of participants
Arm/Group | Magrolimab + Azacitidine | Placebo + Azacitidine
Number analyzed (Participants) | 263 | 264
percentage of participants
  TEAE | 100 | 99.6
  Serious TEAE | 71.9 | 51.5

14. Secondary Outcome: Serum Concentration of Magrolimab
Description: Pretreatment assessments for the initial dose may be collected up to 72 hours before administration of study treatment; thereafter, pretreatment assessments are to be collected within 24 hours prior to study treatment administration.
Time Frame: Preinfusion on Days 0, 7, 28, 56, 112, 168, 252 and 336
Population: Pharmacokinetic (PK) analysis set included all participants who took at least 1 dose of magrolimab and had at least 1 measurable post-treatment serum concentration of magrolimab. Participants with data available at the given timepoint were analyzed.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | Magrolimab + Azacitidine
Number analyzed (Participants) | 218
μg/mL
  Preinfusion Day 0: number analyzed (Participants) | 216
  Preinfusion Day 0 | 0 (0)
  Preinfusion Day 7: number analyzed (Participants) | 205
  Preinfusion Day 7 | 1.09 (15.575)
  Preinfusion Day 28: number analyzed (Participants) | 197
  Preinfusion Day 28 | 500.13 (256.129)
  Preinfusion Day 56: number analyzed (Participants) | 180
  Preinfusion Day 56 | 612.53 (315.037)
  Preinfusion Day 112: number analyzed (Participants) | 125
  Preinfusion Day 112 | 295.64 (178.952)
  Preinfusion Day 168: number analyzed (Participants) | 88
  Preinfusion Day 168 | 258.70 (150.259)
  Preinfusion Day 252: number analyzed (Participants) | 58
  Preinfusion Day 252 | 299.63 (168.944)
  Preinfusion Day 336: number analyzed (Participants) | 42
  Preinfusion Day 336 | 336.57 (241.789)

15. Secondary Outcome: Percentage of Participants With Positive Anti-magrolimab Antibodies
Description: Percentages were rounded off.
Time Frame: Up to 72 hours before administration of any treatment at Day 1, Cycle 1; within 24 hours prior to any study drug administration at Day 1 of Cycles 2, 3, 5, 7, 10, and 13 and End of Treatment (± 7 Days after last study drug dose); Cycle length is 28 Days
Population: Participants in Immunogenicity Analysis Set with at least 1 baseline anti-drug antibody (ADA) sample and at least post-treatment ADA Sample were analyzed. Immunogenicity Analysis Set includes participants who took at least 1 dose of magrolimab and have at least 1 reported ADA result.
Measure: Number; unit: percentage of participants
Arm/Group | Magrolimab + Azacitidine
Number analyzed (Participants) | 230
percentage of participants | 3.5

ADVERSE EVENTS:
Time Frame: Up to 135.9 weeks plus 70 days (Up to 2.8 years)
Description: All cause mortality: The intent-to-treat (ITT) analysis set included all participants who were randomized in the study, with treatment assignments designated according to the treatment that participants were randomized to.
  Adverse Events: The safety analysis set included all randomized participants who received at least 1 dose of any study treatment, with treatment assignments designated according to the actual treatment received.
Arm/Group | Magrolimab + Azacitidine | Placebo + Azacitidine
All-Cause Mortality (participants affected / at risk) | 145/268 | 132/271
Serious Adverse Events (participants affected / at risk) | 189/263 | 136/264
Other Adverse Events (participants affected / at risk) | 246/263 | 256/264
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Magrolimab + Azacitidine (N=263) | Placebo + Azacitidine (N=264)
Anaemia (Blood and lymphatic system disorders) | 25 | 7
Aplastic anaemia (Blood and lymphatic system disorders) | 0 | 1
Cold type haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Extravascular haemolysis (Blood and lymphatic system disorders) | 1 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 2 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 58 | 44
Haemolysis (Blood and lymphatic system disorders) | 9 | 0
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Red blood cell agglutination (Blood and lymphatic system disorders) | 1 | 0
Splenic infarction (Blood and lymphatic system disorders) | 1 | 0
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 6 | 1
Atrial flutter (Cardiac disorders) | 2 | 0
Atrial tachycardia (Cardiac disorders) | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 3 | 4
Cardiac failure (Cardiac disorders) | 4 | 0
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 1 | 1
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Myocarditis (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1
Pulseless electrical activity (Cardiac disorders) | 1 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Stress cardiomyopathy (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 1
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Retinal haemorrhage (Eye disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 3
Anal fistula (Gastrointestinal disorders) | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1
Anal ulcer (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 3
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1
Faecaloma (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 2 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 2
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Mouth swelling (Gastrointestinal disorders) | 0 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 2
Neutropenic colitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 3 | 3
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 5 | 1
Asthenia (General disorders) | 1 | 1
Catheter site haemorrhage (General disorders) | 1 | 0
Chest pain (General disorders) | 3 | 0
Chills (General disorders) | 1 | 0
Death (General disorders) | 1 | 0
Fatigue (General disorders) | 2 | 4
General physical health deterioration (General disorders) | 1 | 0
Generalised oedema (General disorders) | 1 | 0
Hyperthermia (General disorders) | 0 | 1
Influenza like illness (General disorders) | 0 | 1
Injection site irritation (General disorders) | 0 | 1
Localised oedema (General disorders) | 2 | 0
Multiple organ dysfunction syndrome (General disorders) | 2 | 0
Oedema peripheral (General disorders) | 0 | 2
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 17 | 16
Sudden death (General disorders) | 1 | 0
Swelling face (General disorders) | 0 | 1
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Hepatosplenomegaly (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 2 | 0
Hypersensitivity (Immune system disorders) | 1 | 0
Abdominal infection (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1
Arthritis infective (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 5 | 2
Bacterial infection (Infections and infestations) | 0 | 1
Bacterial sepsis (Infections and infestations) | 1 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 2 | 0
Catheter site infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 4 | 7
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 1
Covid-19 (Infections and infestations) | 5 | 10
Covid-19 pneumonia (Infections and infestations) | 1 | 2
Device related infection (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 5 | 1
Empyema (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 2 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Furuncle (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 1 | 0
Hcov-oc43 infection (Infections and infestations) | 1 | 0
Incision site cellulitis (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 1 | 0
Injection site cellulitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lymph node tuberculosis (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 0 | 1
Mucormycosis (Infections and infestations) | 0 | 1
Necrotising fasciitis (Infections and infestations) | 0 | 1
Neutropenic infection (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 6 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 1
Perirectal abscess (Infections and infestations) | 0 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 24 | 11
Pneumonia aspiration (Infections and infestations) | 2 | 1
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pneumonia fungal (Infections and infestations) | 0 | 2
Pneumonia viral (Infections and infestations) | 1 | 1
Post procedural cellulitis (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0
Pseudomonal bacteraemia (Infections and infestations) | 2 | 0
Rash pustular (Infections and infestations) | 1 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 20 | 13
Septic shock (Infections and infestations) | 6 | 4
Sinusitis (Infections and infestations) | 2 | 1
Skin infection (Infections and infestations) | 3 | 2
Soft tissue infection (Infections and infestations) | 1 | 1
Staphylococcal bacteraemia (Infections and infestations) | 1 | 1
Staphylococcal sepsis (Infections and infestations) | 2 | 1
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Thrombophlebitis septic (Infections and infestations) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 7 | 2
Vascular device infection (Infections and infestations) | 3 | 1
Fall (Injury, poisoning and procedural complications) | 3 | 2
Febrile nonhaemolytic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 31 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Synovial rupture (Injury, poisoning and procedural complications) | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 5 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 1 | 1
Vascular procedure complication (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 3 | 0
Amylase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 0
Blood bilirubin increased (Investigations) | 2 | 2
Blood creatinine increased (Investigations) | 1 | 0
Brain natriuretic peptide increased (Investigations) | 1 | 0
Electrocardiogram QT prolonged (Investigations) | 2 | 0
Escherichia test positive (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 1
Oxygen saturation decreased (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 1 | 2
Troponin increased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 1 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle necrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 2 | 1
Dysarthria (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 2 | 1
Facial paralysis (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 2 | 3
Headache (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 1 | 0
Iiird nerve paralysis (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 1
Seizure (Nervous system disorders) | 3 | 1
Sigmoid sinus thrombosis (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 3 | 3
Anxiety (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 2
Delirium (Psychiatric disorders) | 0 | 2
Mental status changes (Psychiatric disorders) | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 4 | 2
Haematuria (Renal and urinary disorders) | 0 | 2
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Urinary bladder haemorrhage (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Balanoposthitis (Reproductive system and breast disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 3
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Blood pressure inadequately controlled (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 2 | 0
Embolism (Vascular disorders) | 2 | 1
Embolism arterial (Vascular disorders) | 1 | 0
Haematoma (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 4 | 6
Orthostatic hypotension (Vascular disorders) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1
Shock haemorrhagic (Vascular disorders) | 2 | 0
Vasculitis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Magrolimab + Azacitidine (N=263) | Placebo + Azacitidine (N=264)
Anaemia (Blood and lymphatic system disorders) | 124 | 75
Febrile neutropenia (Blood and lymphatic system disorders) | 14 | 14
Neutropenia (Blood and lymphatic system disorders) | 63 | 60
Thrombocytopenia (Blood and lymphatic system disorders) | 54 | 46
Atrial fibrillation (Cardiac disorders) | 17 | 9
Palpitations (Cardiac disorders) | 16 | 7
Sinus tachycardia (Cardiac disorders) | 12 | 14
Abdominal pain (Gastrointestinal disorders) | 39 | 25
Constipation (Gastrointestinal disorders) | 144 | 150
Diarrhoea (Gastrointestinal disorders) | 102 | 89
Haemorrhoids (Gastrointestinal disorders) | 13 | 15
Nausea (Gastrointestinal disorders) | 133 | 114
Oral pain (Gastrointestinal disorders) | 17 | 9
Stomatitis (Gastrointestinal disorders) | 22 | 25
Vomiting (Gastrointestinal disorders) | 53 | 55
Asthenia (General disorders) | 22 | 15
Chills (General disorders) | 41 | 22
Fatigue (General disorders) | 105 | 101
Injection site reaction (General disorders) | 18 | 26
Non-cardiac chest pain (General disorders) | 14 | 14
Oedema peripheral (General disorders) | 62 | 46
Pain (General disorders) | 14 | 12
Pyrexia (General disorders) | 75 | 39
Covid-19 (Infections and infestations) | 23 | 22
Pneumonia (Infections and infestations) | 21 | 8
Urinary tract infection (Infections and infestations) | 14 | 13
Contusion (Injury, poisoning and procedural complications) | 31 | 34
Fall (Injury, poisoning and procedural complications) | 29 | 21
Infusion related reaction (Injury, poisoning and procedural complications) | 72 | 40
Alanine aminotransferase increased (Investigations) | 19 | 15
Aspartate aminotransferase increased (Investigations) | 14 | 13
Blood bilirubin increased (Investigations) | 27 | 8
Blood creatinine increased (Investigations) | 13 | 16
Lymphocyte count decreased (Investigations) | 18 | 13
Neutrophil count decreased (Investigations) | 67 | 59
Platelet count decreased (Investigations) | 71 | 64
Weight decreased (Investigations) | 18 | 11
White blood cell count decreased (Investigations) | 47 | 41
Decreased appetite (Metabolism and nutrition disorders) | 72 | 47
Hyperglycaemia (Metabolism and nutrition disorders) | 19 | 15
Hypoalbuminaemia (Metabolism and nutrition disorders) | 20 | 14
Hypokalaemia (Metabolism and nutrition disorders) | 50 | 31
Hypomagnesaemia (Metabolism and nutrition disorders) | 17 | 21
Hyponatraemia (Metabolism and nutrition disorders) | 18 | 18
Hypophosphataemia (Metabolism and nutrition disorders) | 23 | 20
Arthralgia (Musculoskeletal and connective tissue disorders) | 41 | 47
Back pain (Musculoskeletal and connective tissue disorders) | 24 | 21
Muscle spasms (Musculoskeletal and connective tissue disorders) | 13 | 14
Muscular weakness (Musculoskeletal and connective tissue disorders) | 26 | 24
Neck pain (Musculoskeletal and connective tissue disorders) | 6 | 17
Pain in extremity (Musculoskeletal and connective tissue disorders) | 20 | 28
Dizziness (Nervous system disorders) | 46 | 46
Dysgeusia (Nervous system disorders) | 19 | 13
Headache (Nervous system disorders) | 49 | 60
Anxiety (Psychiatric disorders) | 24 | 19
Insomnia (Psychiatric disorders) | 35 | 30
Cough (Respiratory, thoracic and mediastinal disorders) | 55 | 38
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 57 | 42
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 27 | 34
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 14 | 11
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 7 | 16
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 21 | 15
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 20 | 10
Pruritus (Skin and subcutaneous tissue disorders) | 31 | 25
Rash (Skin and subcutaneous tissue disorders) | 19 | 21
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 18 | 16
Hypertension (Vascular disorders) | 16 | 15
Hypotension (Vascular disorders) | 42 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (3):
  • Study Protocol (2022-10-11): https://cdn.clinicaltrials.gov/large-docs/81/NCT04313881/Prot_000.pdf
  • Statistical Analysis Plan: First Interim Analyses (2022-07-29): https://cdn.clinicaltrials.gov/large-docs/81/NCT04313881/SAP_001.pdf
  • Statistical Analysis Plan: Second Interim and Final Analyses (2023-03-06): https://cdn.clinicaltrials.gov/large-docs/81/NCT04313881/SAP_002.pdf